CLINICAL TRIAL: NCT03964129
Title: Clinical Evaluation of Decellularized Nerve Allograft With Autologous Bone Marrow Aspirate Concentrate (BMAC) to Improve Peripheral Nerve Repair and Functional Outcomes
Brief Title: BMAC Nerve Allograft Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency); Curtis National Hand Center at MedStar Union Memorial Hospital (Unknown); Cleveland Clinic Lerner Research Institute (Unknown)
Responsible Party: Principal Investigator, Julia AV Nuelle, Orthopaedic Hand and Microvascular Surgeon, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2017.074
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Nerve Injury Upper Limb

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avance Nerve Graft with autologous BMAC (Experimental): The Avance Nerve Graft will be inserted in the area of nerve injury. Between 40 to 60 ml of Bone Marrow Aspirate from the anterior or posterior iliac crest of the pelvis will be harvested . Using SmartPrep centrifuge and 60 ml BMAC kit, 7 to 10 ml of final BMAC will be obtained.
  Interventions: Procedure: Avance Nerve Graft with Autologous BMAC

INTERVENTIONS:
Procedure: Avance Nerve Graft with Autologous BMAC — The Avance Nerve Graft will be inserted in the area of nerve injury. Between 40 to 60 ml of Bone Marrow Aspirate from the anterior or posterior iliac crest of the pelvis will be harvested. Using SmartPrep centrifuge and 60 ml BMAC kit, 7 to 10 ml of final BMAC will be obtained. Of the 7 to 10 ml of final BMAC that is yielded, half (3.5 to 5 ml) of the final concentrate, will be injected on top of the Avance Nerve Graft following coaptation. The second half (3.5 to 5 ml) of the final concentrate will be inserted into a sterile tube containing culture media and shipped overnight to Cleveland Clinic Lerner Research Institute for cell processing and colony assay to confirm that the BMAC indeed contains autologous bone marrow stem cells.

SUMMARY:
This study is a prospective, multi-center, proof of principle, phase I human safety study evaluating the sequential treatments of the Avance Nerve Graft, a commercially available decellularized processed peripheral nerve allograft, with autologous Bone Marrow Aspirate Concentrate (BMAC), a source of stem cells, for the repair of peripheral nerve injuries up to 7 cm in length. The purpose of this study is to establish a knowledge product, evaluating the safety profile of the Avance Nerve Graft, followed by the application of BMAC to support further investment into the promising area of using stem cells in conjunction with scaffolds.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female 18 to 74 years of age.
* Undergoing peripheral nerve exploration or grafting with allograft in the upper extremity.
* Subjects must be inpatients or scheduled for surgery at the time of study enrollment.
* Has nerve conduction block injuries to the ulnar, median, radial or musculocutaneous nerve of either upper extremities that is less than two years from injury.
* Be willing to undergo tension free end-to-end nerve graft coaptation on both the proximal and distal portion of the nerve gap with the Avance Nerve Graft.
* Be willing to have bone marrow harvested from own body, concentrated, and applied to the site of nerve injury following the insertion of the Avance Nerve Graft.
* Be willing to participate and able to comply with all aspects of the treatment and evaluation schedule over a 18-month duration.
* Capable of giving their own consent to participate in the study, and willing to sign and date an IRB-approved written informed consent prior to initiation of any study procedures.
* Nerve conduction injury affecting sensory and motor function or solely motor function in the upper extremity.
* Nerve gaps following resection, up to 7 cm, inclusive.

Exclusion Criteria:

* Subjects with Type 1 Diabetes Mellitus or Type 2 Diabetes Mellitus requiring regular insulin therapy.
* Subjects who are undergoing or expected to undergo treatment with chemotherapy, radiation therapy, or other known treatment which affects the growth of neural and/or vascular system.
* History of neurodegenerative disease, neuropathy, or diabetic neuropathy.
* History of chronic ischemic condition of the upper extremity.
* Cognitive limitation or mental illness preventing informed consent.
* Nerve injuries >2 years post initial injury.
* Any participant who at the discretion of the Investigator is not suitable for inclusion in the study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the nature and incidence of AEs between the group of subjects receiving Avance Nerve Graft with BMAC and the historical data of nerve repairs with the Avance Nerve Graft. | 18 months
  Long-term study associated AEs, such as infection, wound dehiscence, neuropathy, carpal tunnel syndrome, bleeding, seroma, and lymphocele will be captured and analyzed together with any change in incidence of listed AEs which may be precipitated by treatment. . AEs will be mapped to a MedDRA preferred term and system organ classification. The occurrence of the AEs will be summarized by repair type using MedDRA preferred terms, system organ classifications, and severity. All AEs will be listed for individual subjects showing both verbatim and preferred terms. Separate summaries of treatment-emergent SAEs and AEs related to repair will be generated.

SECONDARY OUTCOMES:
Test of non-inferiority and superiority of Avance Nerve Graft to historical nerve autograft scores with respect to Rosen-Lundborg using closed testing procedures | 18 months
  Test of non-inferiority and superiority of Avance Nerve Graft to historical nerve autograft scores with respect to Rosen-Lundborg will be conducted using closed testing procedures. The hypotheses being tested are as follows:
  H01: Δ ≤ -Δ0 vs. H11: Δ > -Δ0 H02: Δ = 0 vs. H12: Δ ≠ 0 where Δ = μC- μA is the difference between the mean Rosen-Lundborg Scores for the Avance Nerve Graft & BMAC (μA) and the mean Rosen-Lundborg scores for the historical autograft controls (μC), Δ0 is the non-inferiority margin 0.51. The null hypothesis of non-inferiority (H01) will be tested first and, if rejected, then the null hypothesis of superiority (H02) will be assessed. Given that the closed testing procedure is implemented, no adjustment for multiple testing will be required.
Test of non-inferiority of Avance Nerve Graft plus BMAC to Avance Nerve Graft recovery rates with respect to Rosen-Lundborg scores using closed testing procedures | 18 months
  Test of non-inferiority of Avance Nerve Graft plus BMAC to Avance Nerve Graft recovery rates with respect to Rosen-Lundborg scores will be conducted using closed testing procedures. The hypothesis being tested is as follows:
  H01: πA - πAB > Δ vs. H11: πA - πAB < Δ where πA is the recovery of Avance Nerve Graft and πAB is the recovery of Avance plus BMAC. Δ is the non-inferiority margin 25%

OTHER OUTCOMES:
Comparison of Motor Percent Recovery to Baseline Range of Motion | 18 months
  Percent of motor recovery to baseline (defined as the difference in the measured assessment of the repaired nerve as compared with neighboring uninjured and/or contra-lateral side) based on passive range of motion, active range of motion and muscle strength (M0-M5) measurements
Comparison of Motor Percent Recovery to Baseline Grip Strength | 18 months
  Percent of grip strength recovery to baseline (defined as the difference in the measured assessment of the repaired nerve as compared with neighboring uninjured and/or contra-lateral side) measured in kilograms using the Neurosensory & Motor Testing System AcroGrip Device
Comparison of Motor Percent Recovery to Baseline Pinch Strength | 18 months
  Percent of pinch strength recovery to baseline (defined as the difference in the measured assessment of the repaired nerve as compared with neighboring uninjured and/or contra-lateral side) measured in kilograms using the Neurosensory & Motor Testing System AcroPinch Device
Time to Recovery | 18 months
Functional Outcomes through the assessment of Quick Disabilities of the Arm Shoulder and Hand (QuickDASH) questionnaire | 18 months
  QuickDASH Disability/Symptom, Work Module, and Sports/Performing Arts Module Raw Score (out of 5) and Final Score (out of 100) will be recorded. Raw Scores will be calculated by: Raw Score = sum of n responses/n, where n is equal to number of completed items.The Final Score (out of 100) scaled from 0 indicating least disability to 100 indicating most disability will be calculated by: Final score = (Raw Score - 1) X 25
Functional Outcomes through the assessment of Patient-Reported Outcomes Measurement Information System (PROMIS) | 18 months
  Raw and Standardized scores for Physical Function, Pain Intensity, Pain Interference, Fatigue, Sleep Disturbance and Behavior assessments will be recorded. Raw Scores will be calculated by: (Raw Sum X number of items listed in the domain)/Number of items that were actually answered for each assessment. The Raw Score is then systematically transformed to a standardized T-score using a conversion table in the PROMIS Scoring Manual. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. The higher the T-score, the more it represents the concept being measured
Motor and Sensory Nerve Conduction Studies (Nerve Conduction Velocity (NCV) and/or Electromyography (EMG)) | 12 and 18 month
  NCV and EMG testing will be conducted on the target muscle group to assess rate and level of motor and sensory reinnervation in the 12 month and 18 month
  * Rate of Reinnervation (Motor and Sensory Domain)
  * Level of Reinnervation (Motor and Sensory Domain)
Comparison of Sensory Percent Recovery to Baseline | 18 months
  Percent of sensory recovery to baseline (defined as the difference in the measured assessment of the repaired nerve as compared with neighboring uninjured and/or contra-lateral side) using the Neurosensory & Motor Testing System (NSMTS) Pressure Specified Sensory Device. 1 Point Static Discrimination, 1 Point Static Moving Discrimination, 2 Point Static Discrimination and 2 Point Moving Discrimination will be measured by prong pressure (g/mm^2)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Nuelle, MD, Principal Investigator — Brooke Army Medical Center; Leon J Nesti, MD/PhD, Principal Investigator — Walter Reed National Military Medical Center; Kenneth Means, MD, Principal Investigator — Curtis Hand Center at MedStar Union Memorial Hospital
Locations (3):
- United States (3):
  - Curtis National Hand Center at MedStar Union Memorial Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - San Antonio Military Medical Center, Fort Sam Houston, Texas

REFERENCES:
- [Background] Brooks DN, Weber RV, Chao JD, Rinker BD, Zoldos J, Robichaux MR, Ruggeri SB, Anderson KA, Bonatz EE, Wisotsky SM, Cho MS, Wilson C, Cooper EO, Ingari JV, Safa B, Parrett BM, Buncke GM. Processed nerve allografts for peripheral nerve reconstruction: a multicenter study of utilization and outcomes in sensory, mixed, and motor nerve reconstructions. Microsurgery. 2012 Jan;32(1):1-14. doi: 10.1002/micr.20975. Epub 2011 Nov 28. PMID 22121093
- [Background] Berger A, Millesi H. Nerve grafting. Clin Orthop Relat Res. 1978 Jun;(133):49-55. PMID 688717
- [Background] Brushart, T.M. (2011). Nerve Repair (Oxford University Press).
- [Background] Centeno CJ, Al-Sayegh H, Freeman MD, Smith J, Murrell WD, Bubnov R. A multi-center analysis of adverse events among two thousand, three hundred and seventy two adult patients undergoing adult autologous stem cell therapy for orthopaedic conditions. Int Orthop. 2016 Aug;40(8):1755-1765. doi: 10.1007/s00264-016-3162-y. Epub 2016 Mar 30. PMID 27026621
- [Background] Center for Biologics Evaluation and Research, C. for D. and R.H. Cellular & Gene Therapy Guidances - Minimal Manipulation of Human Cells, Tissues, and Cellular and Tissue-Based Products: Draft Guidance.
- [Background] Chen CJ, Ou YC, Liao SL, Chen WY, Chen SY, Wu CW, Wang CC, Wang WY, Huang YS, Hsu SH. Transplantation of bone marrow stromal cells for peripheral nerve repair. Exp Neurol. 2007 Mar;204(1):443-53. doi: 10.1016/j.expneurol.2006.12.004. Epub 2007 Jan 12. PMID 17222827
- [Background] Cho MS, Rinker BD, Weber RV, Chao JD, Ingari JV, Brooks D, Buncke GM. Functional outcome following nerve repair in the upper extremity using processed nerve allograft. J Hand Surg Am. 2012 Nov;37(11):2340-9. doi: 10.1016/j.jhsa.2012.08.028. PMID 23101532
- [Background] Dezawa M, Takahashi I, Esaki M, Takano M, Sawada H. Sciatic nerve regeneration in rats induced by transplantation of in vitro differentiated bone-marrow stromal cells. Eur J Neurosci. 2001 Dec;14(11):1771-6. doi: 10.1046/j.0953-816x.2001.01814.x. PMID 11860471
- [Background] Ding F, Wu J, Yang Y, Hu W, Zhu Q, Tang X, Liu J, Gu X. Use of tissue-engineered nerve grafts consisting of a chitosan/poly(lactic-co-glycolic acid)-based scaffold included with bone marrow mesenchymal cells for bridging 50-mm dog sciatic nerve gaps. Tissue Eng Part A. 2010 Dec;16(12):3779-90. doi: 10.1089/ten.TEA.2010.0299. Epub 2010 Sep 6. PMID 20666610
- [Background] Ducic I, Fu R, Iorio ML. Innovative treatment of peripheral nerve injuries: combined reconstructive concepts. Ann Plast Surg. 2012 Feb;68(2):180-7. doi: 10.1097/SAP.0b013e3182361b23. PMID 22270569
- [Background] Dvali L, Mackinnon S. Nerve repair, grafting, and nerve transfers. Clin Plast Surg. 2003 Apr;30(2):203-21. doi: 10.1016/s0094-1298(02)00096-2. PMID 12737353
- [Background] Frykman, G., and Gramyk, K. (1991). Results of Nerve Grafting In: Gelberman R. Operative nerve repair and reconstruction. (JB Lippincott).
- [Background] Galanakos SP, Zoubos AB, Ignatiadis I, Papakostas I, Gerostathopoulos NE, Soucacos PN. Repair of complete nerve lacerations at the forearm: an outcome study using Rosen-Lundborg protocol. Microsurgery. 2011 May;31(4):253-62. doi: 10.1002/micr.20845. Epub 2010 Dec 3. PMID 21557303
- [Background] Graham, James B., Xue, Qing-Shan, Neubauer, Debbie, and Muir, David (2009). A chondroitinase-treated, decellularized nerve allograft compares favorably to the cellular isograft in rat peripheral nerve repair. 2, 19-29
- [Background] Guo Y, Chen G, Tian G, Tapia C. Sensory recovery following decellularized nerve allograft transplantation for digital nerve repair. J Plast Surg Hand Surg. 2013 Dec;47(6):451-3. doi: 10.3109/2000656X.2013.778862. Epub 2013 Jul 15. PMID 23848418
- [Background] Hegde V, Shonuga O, Ellis S, Fragomen A, Kennedy J, Kudryashov V, Lane JM. A prospective comparison of 3 approved systems for autologous bone marrow concentration demonstrated nonequivalency in progenitor cell number and concentration. J Orthop Trauma. 2014 Oct;28(10):591-8. doi: 10.1097/BOT.0000000000000113. PMID 24694554
- [Background] Hendrich C, Franz E, Waertel G, Krebs R, Jager M. Safety of autologous bone marrow aspiration concentrate transplantation: initial experiences in 101 patients. Orthop Rev (Pavia). 2009 Oct 10;1(2):e32. doi: 10.4081/or.2009.e32. PMID 21808691
- [Background] Hernigou P, Homma Y, Flouzat-Lachaniette CH, Poignard A, Chevallier N, Rouard H. Cancer risk is not increased in patients treated for orthopaedic diseases with autologous bone marrow cell concentrate. J Bone Joint Surg Am. 2013 Dec 18;95(24):2215-21. doi: 10.2106/JBJS.M.00261. PMID 24352775
- [Background] Hu N, Wu H, Xue C, Gong Y, Wu J, Xiao Z, Yang Y, Ding F, Gu X. Long-term outcome of the repair of 50 mm long median nerve defects in rhesus monkeys with marrow mesenchymal stem cells-containing, chitosan-based tissue engineered nerve grafts. Biomaterials. 2013 Jan;34(1):100-11. doi: 10.1016/j.biomaterials.2012.09.020. Epub 2012 Oct 11. PMID 23063298
- [Background] Hu J, Zhu QT, Liu XL, Xu YB, Zhu JK. Repair of extended peripheral nerve lesions in rhesus monkeys using acellular allogenic nerve grafts implanted with autologous mesenchymal stem cells. Exp Neurol. 2007 Apr;204(2):658-66. doi: 10.1016/j.expneurol.2006.11.018. Epub 2007 Jan 10. PMID 17316613
- [Background] IJpma FF, Nicolai JP, Meek MF. Sural nerve donor-site morbidity: thirty-four years of follow-up. Ann Plast Surg. 2006 Oct;57(4):391-5. doi: 10.1097/01.sap.0000221963.66229.b6. PMID 16998330
- [Background] Isaacs J. Major peripheral nerve injuries. Hand Clin. 2013 Aug;29(3):371-82. doi: 10.1016/j.hcl.2013.04.006. Epub 2013 Jun 12. PMID 23895717
- [Background] Jackson WM, Alexander PG, Bulken-Hoover JD, Vogler JA, Ji Y, McKay P, Nesti LJ, Tuan RS. Mesenchymal progenitor cells derived from traumatized muscle enhance neurite growth. J Tissue Eng Regen Med. 2013 Jun;7(6):443-51. doi: 10.1002/term.539. Epub 2012 May 3. PMID 22552971
- [Background] Jager M, Jelinek EM, Wess KM, Scharfstadt A, Jacobson M, Kevy SV, Krauspe R. Bone marrow concentrate: a novel strategy for bone defect treatment. Curr Stem Cell Res Ther. 2009 Jan;4(1):34-43. doi: 10.2174/157488809787169039. PMID 19149628
- [Background] Johnson PJ, Newton P, Hunter DA, Mackinnon SE. Nerve endoneurial microstructure facilitates uniform distribution of regenerative fibers: a post hoc comparison of midgraft nerve fiber densities. J Reconstr Microsurg. 2011 Feb;27(2):83-90. doi: 10.1055/s-0030-1267834. Epub 2010 Oct 13. PMID 20945287
- [Background] Karabekmez FE, Duymaz A, Moran SL. Early clinical outcomes with the use of decellularized nerve allograft for repair of sensory defects within the hand. Hand (N Y). 2009 Sep;4(3):245-9. doi: 10.1007/s11552-009-9195-6. Epub 2009 May 2. PMID 19412640
- [Background] Kragh, Kirby, J.M., and Ficke, J.R. Combat casualty care : lessons learned from OEF and OIF. Chapter 9: Extremity Injury. (2012) Editor-in-chief, Martha K. Lenhart; medical editor, Eric Savitsky; military editor, Brian Eastridge. Pgs. 393-484
- [Background] Lin MY, Manzano G, Gupta R. Nerve allografts and conduits in peripheral nerve repair. Hand Clin. 2013 Aug;29(3):331-48. doi: 10.1016/j.hcl.2013.04.003. PMID 23895714
- [Background] Lohmeyer JA, Siemers F, Machens HG, Mailander P. The clinical use of artificial nerve conduits for digital nerve repair: a prospective cohort study and literature review. J Reconstr Microsurg. 2009 Jan;25(1):55-61. doi: 10.1055/s-0028-1103505. Epub 2008 Nov 26. PMID 19037847
- [Background] Lundborg G. A 25-year perspective of peripheral nerve surgery: evolving neuroscientific concepts and clinical significance. J Hand Surg Am. 2000 May;25(3):391-414. doi: 10.1053/jhsu.2000.4165. PMID 10811744
- [Background] Lundborg G, Rosen B. The two-point discrimination test--time for a re-appraisal? J Hand Surg Br. 2004 Oct;29(5):418-22. doi: 10.1016/j.jhsb.2004.02.008. PMID 15336741
- [Background] Mackinnon SE, Doolabh VB, Novak CB, Trulock EP. Clinical outcome following nerve allograft transplantation. Plast Reconstr Surg. 2001 May;107(6):1419-29. doi: 10.1097/00006534-200105000-00016. PMID 11335811
- [Background] Meek MF, Coert JH, Robinson PH. Poor results after nerve grafting in the upper extremity: Quo vadis? Microsurgery. 2005;25(5):396-402. doi: 10.1002/micr.20137. PMID 16032723
- [Background] Mimura T, Dezawa M, Kanno H, Sawada H, Yamamoto I. Peripheral nerve regeneration by transplantation of bone marrow stromal cell-derived Schwann cells in adult rats. J Neurosurg. 2004 Nov;101(5):806-12. doi: 10.3171/jns.2004.101.5.0806. PMID 15540919
- [Background] Neubauer D, Graham JB, Muir D. Nerve grafts with various sensory and motor fiber compositions are equally effective for the repair of a mixed nerve defect. Exp Neurol. 2010 May;223(1):203-6. doi: 10.1016/j.expneurol.2009.08.013. Epub 2009 Aug 22. PMID 19703442
- [Background] Noble J, Munro CA, Prasad VS, Midha R. Analysis of upper and lower extremity peripheral nerve injuries in a population of patients with multiple injuries. J Trauma. 1998 Jul;45(1):116-22. doi: 10.1097/00005373-199807000-00025. PMID 9680023
- [Background] PRWeb. (2015). AxoGen Inc.'s Avance Nerve Graft Data Presented During Bese Clinical Papers Session at the 70th Annual Meeting of the American Society for Surgery of the Hand. Vocus, Inc. Sep. 10, 2015
- [Background] Reyes M, Verfaillie CM. Characterization of multipotent adult progenitor cells, a subpopulation of mesenchymal stem cells. Ann N Y Acad Sci. 2001 Jun;938:231-3; discussion 233-5. doi: 10.1111/j.1749-6632.2001.tb03593.x. PMID 11458512
- [Background] Rinker B, Liau JY. A prospective randomized study comparing woven polyglycolic acid and autogenous vein conduits for reconstruction of digital nerve gaps. J Hand Surg Am. 2011 May;36(5):775-81. doi: 10.1016/j.jhsa.2011.01.030. Epub 2011 Apr 12. PMID 21489720
- [Background] Siemionow M, Duggan W, Brzezicki G, Klimczak A, Grykien C, Gatherwright J, Nair D. Peripheral nerve defect repair with epineural tubes supported with bone marrow stromal cells: a preliminary report. Ann Plast Surg. 2011 Jul;67(1):73-84. doi: 10.1097/SAP.0b013e318223c2db. PMID 21629045
- [Background] Taras JS, Amin N, Patel N, McCabe LA. Allograft reconstruction for digital nerve loss. J Hand Surg Am. 2013 Oct;38(10):1965-71. doi: 10.1016/j.jhsa.2013.07.008. Epub 2013 Aug 30. PMID 23998191
- [Background] Wakao S, Hayashi T, Kitada M, Kohama M, Matsue D, Teramoto N, Ose T, Itokazu Y, Koshino K, Watabe H, Iida H, Takamoto T, Tabata Y, Dezawa M. Long-term observation of auto-cell transplantation in non-human primate reveals safety and efficiency of bone marrow stromal cell-derived Schwann cells in peripheral nerve regeneration. Exp Neurol. 2010 Jun;223(2):537-47. doi: 10.1016/j.expneurol.2010.01.022. Epub 2010 Feb 11. PMID 20153320
- [Background] Wang D, Liu XL, Zhu JK, Jiang L, Hu J, Zhang Y, Yang LM, Wang HG, Yi JH. Bridging small-gap peripheral nerve defects using acellular nerve allograft implanted with autologous bone marrow stromal cells in primates. Brain Res. 2008 Jan 10;1188:44-53. doi: 10.1016/j.brainres.2007.09.098. Epub 2007 Oct 18. PMID 18061586
- [Background] Wang D, Liu XL, Zhu JK, Hu J, Jiang L, Zhang Y, Yang LM, Wang HG, Zhu QT, Yi JH, Xi TF. Repairing large radial nerve defects by acellular nerve allografts seeded with autologous bone marrow stromal cells in a monkey model. J Neurotrauma. 2010 Oct;27(10):1935-43. doi: 10.1089/neu.2010.1352. PMID 20701436
- [Background] Wangensteen KJ, Kalliainen LK. Collagen tube conduits in peripheral nerve repair: a retrospective analysis. Hand (N Y). 2010 Sep;5(3):273-7. doi: 10.1007/s11552-009-9245-0. Epub 2009 Nov 24. PMID 19937145
- [Background] Weber RA, Breidenbach WC, Brown RE, Jabaley ME, Mass DP. A randomized prospective study of polyglycolic acid conduits for digital nerve reconstruction in humans. Plast Reconstr Surg. 2000 Oct;106(5):1036-45; discussion 1046-8. doi: 10.1097/00006534-200010000-00013. PMID 11039375
- [Background] Whitlock EL, Tuffaha SH, Luciano JP, Yan Y, Hunter DA, Magill CK, Moore AM, Tong AY, Mackinnon SE, Borschel GH. Processed allografts and type I collagen conduits for repair of peripheral nerve gaps. Muscle Nerve. 2009 Jun;39(6):787-99. doi: 10.1002/mus.21220. PMID 19291791
- [Background] Zuniga JR. Sensory outcomes after reconstruction of lingual and inferior alveolar nerve discontinuities using processed nerve allograft--a case series. J Oral Maxillofac Surg. 2015 Apr;73(4):734-44. doi: 10.1016/j.joms.2014.10.030. Epub 2014 Nov 13. PMID 25530279

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT03964129/Prot_SAP_000.pdf